CLINICAL TRIAL: NCT03529331
Title: A Study Comparing Recurrent Use of Morphine Sulfate Immediate Release, Oxycodone/Acetaminophen (Percocet), and Hydrocodone/Acetaminophen (Vicodin) at Discharge From the ED in Opioid-naïve Adult Patients With Moderate to Severe Pain.
Brief Title: A Study Comparing Recurrent Use of MSIR, Percocet, and Vicodin at Discharge From the ED
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The ED physicians no longer prescribe opioids at discharge; not feasible to conduct the study
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-03-01
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: Pain Medications, Analgesia, Emergency Medicine
MeSH Terms: conditions — Pain; Agnosia | interventions — Morphine; oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Morphine Sulfate Immediate Release (Active Comparator): ED patients at discharge will receive 15 mg Morphine Sulfate Immediate Release (MSIR) tablet 4 times a day for 5 days.
  Interventions: Drug: Morphine Sulfate Immediate Release
- Oxycodone/Acetaminophen (Percocet), (Active Comparator): ED patients at discharge will receive 5 mg of Oxycodone/Acetaminophen (Percocet) tablet 4 times a day for 5 days.
  Interventions: Drug: Oxycodone/Acetaminophen
- Hydrocodone/Acetaminophen (Vicodin) (Active Comparator): ED patients at discharge will receive 5 mg of Hydrocodone/Acetaminophen (Vicodin) tablet 4 times a day for 5 days.
  Interventions: Drug: Hydrocodone/Acetaminophen

INTERVENTIONS:
Drug: Morphine Sulfate Immediate Release — 15 mg Morphine Sulfate Immediate Release (MSIR) tablet 4 times a day for 5 days
  Arms: Morphine Sulfate Immediate Release
Drug: Oxycodone/Acetaminophen — 5 mg of Oxycodone/Acetaminophen (Percocet) tablet 4 times a day for 5 days
  Other Names: Percocet
  Arms: Oxycodone/Acetaminophen (Percocet),
Drug: Hydrocodone/Acetaminophen — 5 mg of Hydrocodone/Acetaminophen (Vicodin) tablet 4 times a day for 5 days
  Other Names: Vicodin
  Arms: Hydrocodone/Acetaminophen (Vicodin)

SUMMARY:
This is a prospective randomized, clinical trial comparing recurrent use of Morphine Sulfate Immediate Release (MSIR), Oxycodone/Acetaminophen (Percocet), and Hydrocodone/Acetaminophen (Vicodin) at discharge from the emergency department for opioid-naive adult patients presenting with moderate-to-severe pain. At discharge, patients will be randomized to receive either 5 mg of Oxycodone/Acetaminophen (Percocet) tablet 4 times a day for 5 days, 5 mg of Hydrocodone/Acetaminophen (Vicodin) tablet 4 times a day for 5 days, or 15 mg Morphine Sulfate Immediate Release (MSIR) tablet 4 times a day for 5 days. At 1 month, 3 months, and 6 months patients' prescription's history will be accessed by using the DoctorFirst Drug Database to determine the recurrent use that will serve as a surrogate marker of likeability and abuse liability of each prescribed opioid.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to evaluate and compare rates of recurrent use (surrogate for abuse liability and likeability) of Morphine Sulfate Immediate Release, Oxycodone/Acetaminophen (Percocet), and Hydrocodone/Acetaminophen (Vicodin) at discharge from the ED (by comparing a percentage of patients in each group at 1 month, 3 months and 6 months that are still using the same opioid analgesics for presumably non-medical use.

Objective and Hypothesis:

The outcome of the study is to evaluate and compare the rates of recurrent use of prescribed opioids at discharge from the ED by comparing a percentage of patients in each group at 1 month, 3 months and 6 months that are still using the same opioid analgesics for presumably non-medical use that will be used as a surrogate for comparison of abuse liability and likeability. Our goal is to prove that MSIR will have the lowest recurrent use rates at specified time periods than Percocet and Vicodin and that MSIR should be considered as the opioid of choice at discharge from the ED. Our hypothesis is that MSIR is associated with lower number of patients with recurrent use at specified time periods than Percocet and Vicodin due to the lesser abuse liability and likeability.

Methodology:

This is a prospective randomized, clinical trial comparing recurrent use of Morphine Sulfate Immediate Release (MSIR), Oxycodone/Acetaminophen (Percocet), and Hydrocodone/Acetaminophen (Vicodin) at discharge from the ED for opioid-naive adult patients presenting with moderate-to-severe pain. At discharge, patients will be randomized to receive either 5 mg of Oxycodone/Acetaminophen (Percocet) tablet 4 times a day for 5 days, 5 mg of Hydrocodone/Acetaminophen (Vicodin) tablet 4 times a day for 5 days, or 15 mg Morphine Sulfate Immediate Release (MSIR) tablet 4 times a day for 5 days. At 1 month, 3 months, and 6 months patients' prescription's history will be accessed by using the DoctorFirst Drug Database to determine the recurrent use that will serve as a surrogate marker of likeability and abuse liability of each prescribed opioid.

Statistical Analyses:

The nominal variables will be presented as percentages with confidence intervals (CIs), and continuous variables will be presented as means with SDs, or medians with interquartile ranges when appropriate. The odds ratios of recurrent use will be compared with logistic regression to adjust for age, sex, race, chief complaint, and opioid prescription filling. In addition, to test for proportional difference with respect to recurrent opioid use, we will use a Pearson Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* ED patient
* 18 and older
* acute to moderate to severe pain
* requires oral opioid medications at ED discharge.

Exclusion Criteria:

* chronic non-cancer and cancer pain,
* patients with history of substance abuse
* patients with opioid use disorder,
* patients simultaneously taking antidepressants, benzodiazepines and other sedative-hypnotics,
* and allergies to any of the medications.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients using Prescribed Medication at 1 month | 1 month
  Patients' prescription's history will be accessed by using the DoctorFirst Drug Database to determine the recurrent use that will serve as a surrogate marker of likeability and abuse liability of each prescribed opioid.

SECONDARY OUTCOMES:
Percentage of Patients Using Prescribed Medication at 3 months | 3 months
  Patients' prescription's history will be accessed by using the DoctorFirst Drug Database to determine the recurrent use that will serve as a surrogate marker of likeability and abuse liability of each prescribed opioid.

OTHER OUTCOMES:
Percentage of Patients Using Prescribed Medication at 6 months | 6 months
  Patients' prescription's history will be accessed by using the DoctorFirst Drug Database to determine the recurrent use that will serve as a surrogate marker of likeability and abuse liability of each prescribed opioid.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No